CLINICAL TRIAL: NCT01904279
Title: A Phase Ib, Open-Label, Multicenter Study to Investigate the Pharmacokinetics, Pharmacodynamics, and Safety of Tocilizumab Following Subcutaneous Administration to Patients With Polyarticular Juvenile Idiopathic Arthritis
Brief Title: A Study of Subcutaneously (SC) Administered Tocilizumab (TCZ) in Participants With Polyarticular-Course Juvenile Idiopathic Arthritis (pJIA)
Acronym: JIGSAW 117
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WA28117; 2012-003486-18 (EudraCT Number)
Record Dates: First submitted 2013-06-14; First posted 2013-07-22 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

ARMS (2):
- TCZ SC 162 mg Q3W (Experimental): Participants with body weight less than (<) 30 kilograms (kg) will be administered 162 milligrams (mg) of TCZ as a SC injection every 3 weeks (Q3W) for 52 weeks.
  Interventions: Drug: Tocilizumab
- TCZ SC 162 mg Q2W (Experimental): Participants with body weight greater than or equal to (>/=) 30 kg will be administered 162 mg of TCZ as a SC injection every 2 weeks (Q2W) for 52 weeks.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Participants will receive 162 mg of TCZ as SC injection Q3W or Q2W for 52 weeks
  Other Names: RoActemra/Actemra

SUMMARY:
This open-label, multicenter study evaluated the pharmacokinetics, pharmacodynamics and safety of SC administered TCZ in participants with pJIA.

ELIGIBILITY:
Inclusion Criteria:

* Ages 1 year (12 years for participants in Russia) up to and including 17 years at screening
* Diagnosis of pJIA according to International League of Associations for Rheumatology classification
* Rheumatoid factor (RF)-positive pJIA
* RF-negative pJIA
* Extended oligoarticular JIA with a polyarticular course
* History of inadequate clinical response (in the opinion of the treating physician) to or inability to tolerate methotrexate (MTX)
* Participants currently receiving TCZ by the intravenous (IV) route of administration and with well-controlled disease do not require a period of discontinuation of IV TCZ and should have their first dose of SC TCZ administered on the date that their next IV TCZ infusion would be due. Participants participating in the study may be either naive to TCZ therapy or may be switching from IV to SC. The total number of participants switching from IV TCZ must account for no more than 50 percent (%) of the total participant number. To account for the baseline TCZ concentrations in these participants, information on the last 4 IV TCZ infusions prior to baseline will be collected
* Concurrent treatment with disease-modifying antirheumatic drugs (DMARDs) (including MTX), nonsteroidal anti-inflammatory drugs (NSAIDs), and oral corticosteroids are permitted at the discretion of the investigator
* Females of childbearing potential and non-sterile males with female partner of childbearing potential must agree to use effective contraception as defined by protocol

Exclusion Criteria:

* Prior discontinuation of IV TCZ because of inadequate clinical response or safety events (including hypersensitivity)
* Participants with poorly controlled disease (in the opinion of the treating physician) despite current treatment with IV TCZ
* pJIA that is well controlled by any treatment agent other than TCZ (Juvenile Arthritis Disease Activity Score 71 [JADAS-71] less than or equal to (< / =) 3.8)
* Participants who are wheelchair-bound or bedridden
* Any other auto-immune, rheumatic disease, or overlapping syndrome other than the permitted pcJIA subsets
* Lack of recovery from recent surgery or an interval of <6 weeks since surgery at the time of the screening visit
* Females who are pregnant, lactating, or intending to become pregnant during study conduct
* Any significant concurrent medical or surgical condition that would jeopardize the participant's safety or ability to complete the study
* Known human immunodeficiency virus (HIV) infection or other acquired forms of immune compromise or inborn conditions characterized by a compromised immune system
* History of alcohol, drug, or chemical abuse within 6 months of screening
* Any active acute, subacute, chronic, or recurrent bacterial, viral, or systemic fungal infection or any major episode of infection requiring hospitalization or treatment during screening or treatment with IV antibiotics completed within 4 weeks of the screening visit or oral antibiotics completed within 2 weeks of the screening visit
* History of atypical tuberculosis (TB) or active TB requiring treatment within 2 years prior to screening visit
* Positive purified protein derivative (PPD) at screen, unless treated with anti-TB therapy for at least 4 weeks prior to receiving study drug and chest radiograph is negative for active TB within 6 months of screening visit according to local practice
* History of reactivation or new onset of a systemic infection such as herpes zoster or Epstein-Barr virus within 2 months of the screening visit
* Hepatitis B surface antigen or hepatitis C antibody positivity or chronic viral or autoimmune hepatitis
* History of concurrent serious gastrointestinal disorders such as ulcer or inflammatory bowel disease, Crohn's disease, ulcerative colitis, or other symptomatic lower gastrointestinal conditions
* History of or current cancer or lymphoma
* Uncontrolled diabetes mellitus with elevated glycosylated hemoglobin
* Active uveitis at screening
* Inadequate hematologic, renal or liver function
* Prior stem cell transplant at any time

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2013-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- United States (9):
  - Hartford, Connecticut
  - Chicago, Illinois
  - Hackensack, New Jersey
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Tulsa, Oklahoma
  - Salt Lake City, Utah
  - Seattle, Washington
- Buenos Aires, Argentina
- Australia (2):
  - Westmead, New South Wales
  - Parkville, Victoria
- Brazil (2):
  - Rio de Janeiro, Rio de Janeiro
  - São Paulo, São Paulo
- Canada (3):
  - Calgary, Alberta
  - Ottawa, Ontario
  - Toronto, Ontario
- Le Kremlin-Bicêtre, France
- Germany (3):
  - Berlin
  - Freiburg im Breisgau
  - Sankt Augustin
- Italy (3):
  - Rome, Lazio
  - Genoa, Liguria
  - Florence, Tuscany
- Monterrey, Mexico
- Moscow, Russia
- Spain (2):
  - Esplugas de Llobregat, Barcelona
  - Madrid
- United Kingdom (2):
  - Bristol
  - Liverpool

REFERENCES:
- [Derived] Ruperto N, Brunner HI, Ramanan AV, Horneff G, Cuttica R, Henrickson M, Anton J, Boteanu AL, Penades IC, Minden K, Schmeling H, Hufnagel M, Weiss JE, Pardeo M, Nanda K, Roth J, Rubio-Perez N, Hsu JC, Wimalasundera S, Wells C, Bharucha K, Douglass W, Bao M, Mallalieu NL, Martini A, Lovell D, Benedetti F; Paediatric Rheumatology INternational Trials Organisation (PRINTO) and the Paediatric Rheumatology Collaborative Study Group (PRCSG). Subcutaneous dosing regimens of tocilizumab in children with systemic or polyarticular juvenile idiopathic arthritis. Rheumatology (Oxford). 2021 Oct 2;60(10):4568-4580. doi: 10.1093/rheumatology/keab047. PMID 33506875

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 52 participants were enrolled in the study. Study included a 21-day screening period.
Groups:
- TCZ SC 162 mg Q3W: Participants with body weight less than (<) 30 kilograms (kg) were administered 162 milligrams (mg) of TCZ as an subcutaneous (SC) injection every 3 weeks (Q3W) for 52 weeks.
- TCZ SC 162 mg Q2W: Participants with body weight greater than or equal to (>/=) 30 kg were administered 162 mg of TCZ as an SC injection every 2 weeks (Q2W) for 52 weeks.
Period: Overall Study
Arm/Group | TCZ SC 162 mg Q3W | TCZ SC 162 mg Q2W
Started | 27 | 25
Completed | 24 | 22
Not Completed | 3 | 3
Not completed — Lack of Efficacy | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of treatment and who had at least one post-dose safety assessment.
Groups:
- TCZ SC 162 mg Q3W: Participants with body weight < 30 kg were administered 162 mg of TCZ as an SC injection Q3W for 52 weeks.
- TCZ SC 162 mg Q2W: Participants with body weight >/= 30 kg were administered 162 mg of TCZ as an SC injection Q2W for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | TCZ SC 162 mg Q3W | TCZ SC 162 mg Q2W | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.5 (2.1) | 13.9 (2.7) | 9.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Minimum Serum Concentration (Cmin) of TCZ at Steady State
Description: Detailed timeframe for TCZ SC 162 mg Q3W arm: pre-dose (Hour 0), 96, 504, 1008, 2016, 2022, 2064, 2112, 2160, 2520 hours post Day 1 dose (additionally at 6, 12, 48, 120, 2028 hours post Day 1 dose in participants >/=2 years old). Detailed timeframe for TCZ SC 162 mg Q2W arm: pre-dose (Hour 0), 6, 12, 48, 120, 336, 672, 1008, 2016, 2022, 2028, 2040, 2064, 2112, 2160, 2520 hours post Day 1 dose.
Time Frame: Pre-dose (Hour 0) up to 2520 hours post Day 1 dose (detailed timeframe is provided in outcome description section)
Population: Pharmacokinetic population included all enrolled participants who were adherent to the protocol.
Measure: Median (Full Range); unit: Micrograms/milliliter (mcg/mL)
Arm/Group | TCZ SC 162 mg Q3W | TCZ SC 162 mg Q2W
Number analyzed (Participants) | 27 | 25
Micrograms/milliliter (mcg/mL) | 13.35 [0.21 to 52.25] | 12.71 [0.19 to 23.75]

2. Primary Outcome: Area Under the Curve at Steady-state Over a 12-week Interval (AUC12weeks) of TCZ Treatment
Description: Detailed timeframe for TCZ SC 162 mg Q3W arm: pre-dose (Hour 0), 96, 504, 1008, 2016 hours post Day 1 dose (additionally at 6, 12, 48, 120 hours post Day 1 dose in participants >/=2 years old). Detailed timeframe for TCZ SC 162 mg Q2W arm: pre-dose (Hour 0), 6, 12, 48, 120, 336, 672, 1008, 2016 post Day 1 dose.
Time Frame: Pre-dose (Hour 0) up to 2016 hours post Day 1 dose (detailed timeframe is provided in outcome description section)
Population: Pharmacokinetic population.
Measure: Mean (Full Range); unit: mcg*day/mL
Arm/Group | TCZ SC 162 mg Q3W | TCZ SC 162 mg Q2W
Number analyzed (Participants) | 27 | 25
mcg*day/mL | 2998 [1465 to 7708] | 1933 [324 to 3098]

3. Primary Outcome: Maximum Serum Concentration (Cmax) of TCZ at Steady State
Description: Detailed timeframe for TCZ SC 162 mg Q3W arm: pre-dose (Hour 0), 96, 504, 1008, 2016, 2022, 2064, 2112, ,2160, 2520 hours post Day 1 dose (additionally at 6, 12, 48, 120, 2028 hours post Day 1 dose in participants >/=2 years old). Detailed timeframe for TCZ SC 162 mg Q2W arm: pre-dose (Hour 0), 6, 12, 48, 120, 336, 672, 1008, 2016, 2022, 2028, 2040, 2064, 2112, 2160, 2520 hours post Day 1 dose.
Time Frame: Pre-dose (Hour 0) up to 2520 hours post Day 1 dose (detailed timeframe is provided in outcome description section)
Population: Pharmacokinetic population
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | TCZ SC 162 mg Q3W | TCZ SC 162 mg Q2W
Number analyzed (Participants) | 27 | 25
mcg/mL | 62.44 [39.37 to 121.13] | 29.74 [7.56 to 50.3]

4. Secondary Outcome: Change From Baseline in Serum Interleukin-6 (IL-6) Levels
Description: IL-6 is a cytokine associated with disease activity in juvenile idiopathic arthritis (JIA) including the polyarticular juvenile idiopathic arthritis (pJIA) subset. It is found in high levels in the synovial fluid and is associated with indicators of inflammatory activity.
Time Frame: Baseline, Days 0.25, 0.5, 2, 4, 5, 84.25, 84.5, 85, 86, 88, 90; Weeks 2, 3, 4, 6, 12, 14, 15, 27, 28, 36, 44, 52
Population: Safety population. Here Number of participants analyzed represents participants evaluable for this outcome measure. Number Analyzed represents participants evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: picograms/milliliter (pg/mL)
Arm/Group | TCZ SC 162 mg Q3W | TCZ SC 162 mg Q2W
Number analyzed (Participants) | 18 | 23
picograms/milliliter (pg/mL)
  Baseline | 77.569 (278.376) | 10.567 (11.24)
  Day 0.25 | -15.309 (108.157) | 4.575 (7.555)
  Day 0.5: number analyzed (Participants) | 15 | 23
  Day 0.5 | -16.181 (116.587) | 11.932 (13.33)
  Day 2 | 17.998 (157.295) | 23.223 (23.935)
  Day 4: number analyzed (Participants) | 0 | 0
  Day 5: number analyzed (Participants) | 17 | 23
  Day 5 | 17.265 (186.212) | 35.263 (64.907)
  Week 2: number analyzed (Participants) | 0 | 23
  Week 2 |  | 21.751 (49.964)
  Week 3: number analyzed (Participants) | 18 | 0
  Week 3 | -12.801 (198.038) |
  Week 4: number analyzed (Participants) | 0 | 22
  Week 4 |  | 15.944 (26.322)
  Week 6 | -0.412 (271.409) | 17.841 (34.515)
  Week 12: number analyzed (Participants) | 16 | 21
  Week 12 | -45.569 (294.169) | 17.236 (28.727)
  Day 84.25: number analyzed (Participants) | 14 | 21
  Day 84.25 | 32.644 (65.094) | 14.66 (24.026)
  Day 84.5: number analyzed (Participants) | 13 | 20
  Day 84.5 | -46.575 (318.217) | 24.478 (31.747)
  Day 85: number analyzed (Participants) | 0 | 22
  Day 85 |  | 27.934 (53.23)
  Day 86: number analyzed (Participants) | 16 | 21
  Day 86 | -53.35 (285.831) | 36.06 (82.547)
  Day 88: number analyzed (Participants) | 17 | 21
  Day 88 | -42.836 (280.041) | 19.397 (22.712)
  Day 90: number analyzed (Participants) | 15 | 19
  Day 90 | -51.899 (299.59) | 20.642 (20.247)
  Week 14: number analyzed (Participants) | 0 | 23
  Week 14 |  | 11.958 (16.665)
  Week 15: number analyzed (Participants) | 17 | 1
  Week 15 | -21.565 (312.758) | 122.88
  Week 27: number analyzed (Participants) | 18 | 0
  Week 27 | -16.408 (293.156) |
  Week 28: number analyzed (Participants) | 0 | 20
  Week 28 |  | 14.206 (20.762)
  Week 36: number analyzed (Participants) | 16 | 16
  Week 36 | -38.921 (303.851) | 13.273 (24.814)
  Week 44: number analyzed (Participants) | 0 | 20
  Week 44 |  | 14.765 (18.458)
  Week 52: number analyzed (Participants) | 17 | 20
  Week 52 | -44.611 (289.698) | 10.401 (18.455)

5. Secondary Outcome: Change From Baseline in Soluble IL-6 Receptor Levels
Time Frame: Baseline, Days 0.25, 0.5, 2, 4, 5, 84.25, 84.5, 85, 86, 88, 90; Weeks 2, 3, 4, 6, 12, 14, 15, 27, 28, 36, 44, 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | TCZ SC 162 mg Q3W | TCZ SC 162 mg Q2W
Number analyzed (Participants) | 20 | 23
nanograms per milliliter (ng/mL)
  Baseline | 140.4 (225.72) | 206.7 (241.69)
  Day 0.25: number analyzed (Participants) | 19 | 23
  Day 0.25 | -4.04 (41.14) | 1.78 (29.68)
  Day 0.5: number analyzed (Participants) | 16 | 22
  Day 0.5 | -1.45 (53.39) | 4.58 (51.71)
  Day 2: number analyzed (Participants) | 19 | 23
  Day 2 | 89.72 (75.29) | 68.90 (66.75)
  Day 4: number analyzed (Participants) | 1 | 0
  Day 4 | 323.4 (NA) — The data was not available as single participant was evaluated. |
  Day 5: number analyzed (Participants) | 19 | 23
  Day 5 | 194.46 (143.28) | 124.65 (100.58)
  Week 2: number analyzed (Participants) | 0 | 23
  Week 2 |  | 193.25 (158.69)
  Week 3: number analyzed (Participants) | 20 | 0
  Week 3 | 418.54 (237.02) |
  Week 4: number analyzed (Participants) | 0 | 23
  Week 4 |  | 239.86 (194.47)
  Week 6 | 407.36 (344.44) | 233.82 (234.92)
  Week 12: number analyzed (Participants) | 17 | 21
  Week 12 | 464.77 (317.77) | 286.06 (260.33)
  Day 84.25: number analyzed (Participants) | 17 | 23
  Day 84.25 | 461.85 (280.99) | 245.05 (253.45)
  Day 84.5: number analyzed (Participants) | 17 | 22
  Day 84.5 | 482.55 (299.43) | 274.85 (230.86)
  Day 85: number analyzed (Participants) | 0 | 22
  Day 85 |  | 268.72 (254.46)
  Day 86: number analyzed (Participants) | 19 | 22
  Day 86 | 461.19 (345.97) | 244.53 (257.08)
  Day 88: number analyzed (Participants) | 19 | 21
  Day 88 | 514.89 (303.29) | 256.47 (234.7)
  Day 90: number analyzed (Participants) | 19 | 20
  Day 90 | 494.05 (276.35) | 292.29 (229.2)
  Week 14: number analyzed (Participants) | 0 | 23
  Week 14 |  | 272.93 (241.9)
  Week 15: number analyzed (Participants) | 20 | 1
  Week 15 | 497.21 (295.29) | 200 (NA) — The data was not available as single participant was evaluated.
  Week 27: number analyzed (Participants) | 20 | 0
  Week 27 | 532.81 (270.07) |
  Week 28: number analyzed (Participants) | 0 | 21
  Week 28 |  | 295.28 (286.78)
  Week 36: number analyzed (Participants) | 18 | 18
  Week 36 | 416.02 (305.07) | 269.32 (276.03)
  Week 44: number analyzed (Participants) | 0 | 21
  Week 44 |  | 243.93 (299.72)
  Week 52: number analyzed (Participants) | 20 | 22
  Week 52 | 470.6 (263.38) | 209.51 (318.38)

6. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) Levels
Time Frame: Baseline, Weeks 4, 6, 9, 12,18, 20, 27, 28, 36, 44, 45, 51, 52
Population: Safety population. Number Analyzed represents participants evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | TCZ SC 162 mg Q3W | TCZ SC 162 mg Q2W
Number analyzed (Participants) | 27 | 25
mg/L
  Baseline | 3.391 (5.27) | 3.356 (6.908)
  Week 4: number analyzed (Participants) | 0 | 25
  Week 4 |  | -2.187 (5.270)
  Week 6 | -3 (5.21) | -2.368 (5.735)
  Week 9: number analyzed (Participants) | 27 | 0
  Week 9 | -3.069 (5.346) |
  Week 12: number analyzed (Participants) | 27 | 24
  Week 12 | -3.16 (5.285) | -1.783 (4.559)
  Week 18: number analyzed (Participants) | 26 | 0
  Week 18 | -3.213 (5.377) |
  Week 20: number analyzed (Participants) | 0 | 25
  Week 20 |  | -1.336 (6.158)
  Week 27: number analyzed (Participants) | 27 | 0
  Week 27 | -3.122 (5.279) |
  Week 28: number analyzed (Participants) | 0 | 25
  Week 28 |  | -2.467 (6.455)
  Week 36: number analyzed (Participants) | 25 | 22
  Week 36 | -3.254 (5.492) | -2.209 (5.316)
  Week 44: number analyzed (Participants) | 0 | 22
  Week 44 |  | -2.039 (5.47)
  Week 45: number analyzed (Participants) | 26 | 0
  Week 45 | -3.153 (5.385) |
  Week 51: number analyzed (Participants) | 25 | 0
  Week 51 | -3.344 (5.453) |
  Week 52: number analyzed (Participants) | 0 | 22
  Week 52 |  | -2.225 (5.285)

7. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: The ESR is an acute phase reactant and a measure of inflammation. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 4, 6, 9, 12, 18, 20, 27, 28, 36, 44, 45, 51, 52
Population: Safety population. Number Analyzed represents participants evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: millimeters per hour (mm/h)
Arm/Group | TCZ SC 162 mg Q3W | TCZ SC 162 mg Q2W
Number analyzed (Participants) | 27 | 25
millimeters per hour (mm/h)
  Baseline | 15.9 (14.2) | 13 (13.1)
  Week 4: number analyzed (Participants) | 0 | 25
  Week 4 |  | -7.0 (9)
  Week 6: number analyzed (Participants) | 26 | 25
  Week 6 | -10.6 (12.8) | -7.2 (10.5)
  Week 9: number analyzed (Participants) | 25 | 0
  Week 9 | -9.9 (10.9) |
  Week 12: number analyzed (Participants) | 26 | 25
  Week 12 | -9.8 (12.4) | -6.8 (13)
  Week 18: number analyzed (Participants) | 26 | 0
  Week 18 | -11.8 (12.3) |
  Week 20: number analyzed (Participants) | 0 | 25
  Week 20 |  | -7.9 (11.2)
  Week 27: number analyzed (Participants) | 27 | 0
  Week 27 | -11.9 (12.2) |
  Week 28: number analyzed (Participants) | 0 | 23
  Week 28 |  | -8 (14.2)
  Week 36: number analyzed (Participants) | 26 | 21
  Week 36 | -11.8 (12.8) | -8 (13.1)
  Week 44: number analyzed (Participants) | 0 | 21
  Week 44 |  | -10.2 (13)
  Week 45: number analyzed (Participants) | 26 | 0
  Week 45 | -12 (12.2) |
  Week 51: number analyzed (Participants) | 25 | 0
  Week 51 | -12.2 (13) |
  Week 52: number analyzed (Participants) | 0 | 22
  Week 52 |  | -8.5 (13.2)

8. Secondary Outcome: Percentage of Participants With Anti-TCZ Antibodies of Neutralizing Potential
Time Frame: Baseline up to Week 52
Population: Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | TCZ SC 162 mg Q3W | TCZ SC 162 mg Q2W
Number analyzed (Participants) | 27 | 25
percentage of participants | 3.7 | 8.0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 56
Description: Safety population
Arm/Group | TCZ SC 162 mg Q3W | TCZ SC 162 mg Q2W
Serious Adverse Events (participants affected / at risk) | 1/27 | 2/25
Other Adverse Events (participants affected / at risk) | 23/27 | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TCZ SC 162 mg Q3W (N=27) | TCZ SC 162 mg Q2W (N=25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Croup infectious (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TCZ SC 162 mg Q3W (N=27) | TCZ SC 162 mg Q2W (N=25)
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Ear Pain (Ear and labyrinth disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 3
Aphthous Ulcer (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 1 | 5
Vomiting (Gastrointestinal disorders) | 4 | 5
Fatigue (General disorders) | 0 | 2
Injection Site Erythema (General disorders) | 4 | 6
Injection Site Haematoma (General disorders) | 0 | 2
Injection Site Pain (General disorders) | 0 | 2
Injection Site Pruritus (General disorders) | 0 | 2
Injection Site Swelling (General disorders) | 1 | 2
Pyrexia (General disorders) | 2 | 4
Vessel Puncture Site Haematoma (General disorders) | 0 | 2
Bronchitis (Infections and infestations) | 2 | 1
Ear Infection (Infections and infestations) | 4 | 0
Gastroenteritis (Infections and infestations) | 4 | 2
Impetigo (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 2 | 0
Nasophryngitis (Infections and infestations) | 11 | 7
Otitis Media (Infections and infestations) | 3 | 0
Paronychia (Infections and infestations) | 0 | 2
Rhinitis (Infections and infestations) | 1 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 4
Viral Infection (Infections and infestations) | 2 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Juvenile Idiopathic Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Headache (Nervous system disorders) | 1 | 6
Insomnia (Psychiatric disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Haematoma (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.